CLINICAL TRIAL: NCT00463177
Title: Augmented Cerebral Pain Processing in Chronic, Unexplained Pain: a 3T Event-Related Functional MRI Study
Brief Title: Augmented Cerebral Pain Processing in Chronic, Unexplained Pain: a fMRI Study
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: K.F. Hein Foundation (Other); Fonds Psychische Gezondheid (Other)
Responsible Party: UMC Utrecht
Other Study IDs: NFGV5503-02
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Pain
Keywords: Pain; Chronic pain; Pain disorder; Functional MRI; Sensitization
MeSH Terms: conditions — Pain; Chronic Pain; Somatoform Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic, unexplained pain symptoms are very common in all layers of the population, but it is largely unknown what causes them. This study examines the hypothesis that patients with these pain symptoms process pain abnormally in their brain. TO this aim, we compare patients and healthy people: they receive mild pain at their painful body region and at another location. Concurrently, we measure brain activity with brain scans (functional MRI scans). With our study results, we want to increase understanding of what causes chronic, unexplained pain symptoms, in order to find better methods of diagnosing and treating them.

DETAILED DESCRIPTION:
Background

Chronic, unexplained pain is a heterogeneously defined, but common and recurring clinical problem, in general medical practice as well as in specialist care. Chronic, unexplained pain causes considerable loss of quality of life, frequent absence from work and it is a common reason for health care visits. From a pathophysiological point of view, an augmented and self-amplifying sensitivity for physical signals such as pain (as well as for other signals) seems to be important. This is referred to as 'generalised hypervigilance', a specific type of sensitisation. Central sensitisation mechanisms have been implied in several pain syndromes. In our own psychophysical pilot study, we confirmed the existence of amplified pain perception in chronic, unexplained pain, as well as the disturbed influence of attentional processes. Our study results probably reflect a general disturbance of perception, not associated with a specific body location. This general perceptual disturbance is expressed in a stronger fashion in the clinically affected body region. Abnormal pattern of cerebral pain processing have been found in functional MRI studies in other syndromes of unknown origin, such as fibromyalgia, somatoform pain disorder and irritable bowel syndrome. However, the role of several neurobiological factors in chronic, unexplained pain remain to be elucidated and to be placed in the context of the biopsychosocial model.

Work plan:

A 3T rapid event-related, Functional MRI-experiment into the cerebral processing of experimental pain stimuli in chronic, unexplained pain-patients versus healthy controls. Twelve chronic, unexplained pain-patients with unilateral limb pain and twelve healthy control subjects experience painful and non-painful electrical stimuli on the painful limb, whilst the attentional state of the subject is controlled. With functional MRI, we record the pain-related cerebral activations and compare them between groups, in order to characterise the cerebral correlates of altered pain processing in chronic, unexplained pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic limb pain > 6 months
* No known somatic cause

Exclusion Criteria:

* Chronic benzodiazepine use
* Axis-I psychiatric co-morbidity
* Contra-indications for MRI scanning (e.g. implanted pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic unexplained pain patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Snijders, MD, Principal Investigator — UMC Utrecht; Jan van Gijn, MD, Study Chair — UMC Utrecht; Nick Ramsey, PhD, Study Director — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands